CLINICAL TRIAL: NCT02809976
Title: Open Label Phase 2 Proof-of-concept Pilot Trial of Topical Ruxolitinib in Repigmenting Adult Patients With Vitiligo
Brief Title: Topical Ruxolitinib for the Treatment of Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-18424-15-06
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib 1.5% phosphate cream (Experimental): Ruxolitinib 1.5% phosphate cream twice daily to vitiligo patches.
  Interventions: Drug: Ruxolitinib 1.5% Phosphate Cream

INTERVENTIONS:
Drug: Ruxolitinib 1.5% Phosphate Cream — twice daily topical application of Ruxolitinib 1.5% Phosphate Cream beginning at baseline and ending at week 20
  Other Names: INCB018424 phosphate cream

SUMMARY:
The purpose of this study is to determine if topical ruxolitinib 1.5% will provide repigmentation in vitiligo lesions.

DETAILED DESCRIPTION:
The hypothesis is that JAK inhibitors can also successfully treat vitiligo. Lesional skin of both alopecia areata and vitiligo primarily contain T cells in a TH1 response as opposed to a mixed cell infiltrate such as in psoriasis or lichen planus. Both alopecia areata and vitiligo are TH1 mediated diseases dependent on the production of IFN-gamma to drive the response. CD8+ T cells are both necessary and sufficient for melanocyte destruction in vitiligo (van den Boorn JG et al 2009) and CD8+NKG2D+ T cells are also necessary and sufficient for hair loss in alopecia areata (Gilhar A et al 2013).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of vitiligo.
* At Visit 1 (Baseline/Day 1), have had vitiligo covering at least 1% of total body surface area (BSA) on the scalp, trunk or limbs (excluding nails).
* Female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least four weeks after the last dose of assigned treatment. Male subjects must also use contraception, such as barrier method with spermicide.
* If receiving concomitant medications for any reason, must be on a stable regimen and willing to stay on a stable regimen.
* Must be willing to washout of other vitiligo treatments. All treatments for vitiligo are prohibited during the course of the study.

Exclusion Criteria:

* Other skin conditions at Baseline that would interfere with evaluation of vitiligo.
* Pregnant/breastfeeding females, or females of childbearing potential not using highly effective contraception. Women of childbearing potential must test negative for pregnancy and use contraception for at least four weeks after last dose of drug.
* Current or recent history of clinically significant medical/psychiatric condition or laboratory abnormality that may increase risk associated with the study participation or drug administration.
* Have a history of any lymphoproliferative disorder, lymphoma, leukemia, history of disseminated herpes zoster or disseminated herpes simplex, or a recurrent localized, dermatomal herpes zoster.
* Have a history of infection requiring parenteral or oral or topical antimicrobial therapy within 2 weeks prior to Baseline.
* Vaccinated with live/attenuated live vaccine within 6 weeks prior to Baseline.
* Previously participated in study of oral/topical ruxolitinib or tofacitinib (tofacitinib, CP-690,550, formerly tasocitinib) unless confirmed to have been randomized to and treated with placebo or placebo topical formulation (vehicle) only.
* Received a prohibited concomitant medication within 7 days or 5 half-lives (whichever is longer) prior to Baseline.
* Have participated in other studies within 4 weeks or 5 half-lives (whichever is longer) prior to Visit 1 (Baseline/Day 1). Subjects cannot participate in studies of other investigational or experimental therapies or procedures at any time during their participation in this study.
* Subjects who are investigational site staff members or relatives of those site staff members or subjects who are Sponsor employees directly involved in the conduct of the trial.
* In the opinion of the investigator or Sponsor, the subject is inappropriate for entry into this study, or unwilling/unable to comply with study procedures and lifestyle guidelines.
* Screening laboratory abnormalities
* CYP Inhibitor Exclusion: Subjects taking potent CYP3A4 inhibitors or fluconazole within 2 weeks or 5 half-lives, whichever is longer, before the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rosmarin, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Started | 11
Completed | 9
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 52 [33 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Vitiligo Area Severity Index (VASI) Score From Baseline to Week 20
Description: The VASI for each body region (hands, upper extremities, trunk, lower extremities, feet) is determined by the product of the area involved in hand prints and the extent of depigmentation within each hand print unit measured patch (0-100). Area involved is measured by hand prints (1 hand print = 1%) with a possible range of 0-100. Degree of depigmentation is measured as: 1.00 (100%) = complete depigmentation, no pigment present, 0.90(90%)=specks of pigment present, 0.75(75%)=depigmented area exceeds the pigmented area, 0.50(50%)=pigmented and depigmented areas are equal, 0.25(25%)=pigmented area exceeds depigmented area, 0.10(10%)=only specks of depigmentation present, and 0.0(0%)=no depigmentation present.
Time Frame: Baseline to Week 20
Measure: Mean (95% Confidence Interval); unit: percentage of change in VASI
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
percentage of change in VASI | 23 [4 to 43]
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Phosphate Cream; Test type: Other — single group/descriptive analysis; p = 0.02, paired t-test

2. Secondary Outcome: Percent Change in Body Surface Area (BSA) of Repigmentation
Description: Area involved is measured by hand prints (1 hand print = 1%) with a possible range of 0-100.
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
percentage of change | 11.2 (26.4)

3. Secondary Outcome: Number of Subjects Who Achieve a Physician Global Vitiligo Assessment (PGVA) of Clear or Almost Clear
Time Frame: Baseline and Week 20
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
Participants | 2

4. Secondary Outcome: Percent Change in Vitiligo European Task Force (VETF) Assessment - Body Surface Area
Description: Vitiligo European Task Force assessment consisted of three components: Extent of disease reflecting the body surface area (0-100%), disease staging (0-20), and disease progression (-5 +5). Staging is based on cutaneous and hair pigmentation assessing the largest patch in each body area (head/neck, trunk, arms, legs, and hands/feet); Stage 0=normal pigmentation, Stage 1=incomplete pigmentation, Stage 2=complete depigmentation, Stage 3= partial hair whitening (<30%), Stage 4= complete hair whitening. Disease progression is based on assessing the largest patch in each body area; Score 0= similar limits, Score 1= progressive vitiligo (ongoing subclinical depigmentation), Score -1= regressive vitiligo (ongoing subclinical repigmentation). Where a higher number indicates more severe disease spread and a negative number indicates improving disease. These three subsets are evaluated and reported independently and not mutually related to each other.
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: percent change in body surface area
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
percent change in body surface area | 11.2 (26.4)

5. Secondary Outcome: Mean Dermatology Life Quality Index (DLQI) Scores
Description: DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The percent change was calculated from the mean DLQI at baseline and week 20
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
score on a scale
  Week 20 | 3 (3.46)
  Baseline | 2.9 (2.67)

6. Secondary Outcome: Percent Change in Vitiligo European Task Force (VETF) Assessment - Disease Staging
Description: as for outcome 4
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: percent change in disease staging score
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
percent change in disease staging score | 4.5 (2.4)

7. Secondary Outcome: Percent Change in Vitiligo European Task Force (VETF) Assessment - Disease Progression
Description: as for outcome 4
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: percent of change
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
Number analyzed (Participants) | 11
percent of change | -0.5 (1.1)

ADVERSE EVENTS:
Arm/Group | Ruxolitinib 1.5% Phosphate Cream
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib 1.5% Phosphate Cream (N=11)
Rim of hyperpigmentation surrounding vitiligo lesion (Skin and subcutaneous tissue disorders) | 9
Intermittent erythema over affected lesions (Skin and subcutaneous tissue disorders) | 8
Transient acne (Skin and subcutaneous tissue disorders) | 2
URI symptoms (Respiratory, thoracic and mediastinal disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Muscle aches (Musculoskeletal and connective tissue disorders) | 1
hypercholesterolemia (Metabolism and nutrition disorders) | 1
Traumatic blister (Social circumstances) | 1
Bee sting (Social circumstances) | 1
Dental pain (General disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No